CLINICAL TRIAL: NCT01719978
Title: Hemodynamic and Electrocardiographic Effects of Hyaluronidase Associated With Local Anaesthetics: a Double-blind "Split-mouth" Controlled Trial.
Brief Title: Hemodynamic and Electrocardiographic Effects of Hyaluronidase Associated With Local Anaesthetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mauricio Jose Tornelli (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor-Investigator, Mauricio Jose Tornelli, PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MTornelli
Record Dates: First submitted 2012-10-03; First posted 2012-11-01 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Cardiac Arrhythmias
Keywords: Local Anaesthetics; Mepivacaine; hyaluronoglucosaminidase; Hemodynamic; Electrocardiography and Dentistry.
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Mepivacaine; Epinephrine; Hyaluronoglucosaminidase; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronidase (Active Comparator): Lower Third Molar Extraction -- 3.6mL 2% Mepivacaine with 1:100,000 epinephrine + Hyaluronidase
  Interventions: Drug: 3.6mL 2% Mepivacaine with 1:100,000 epinephrine; Procedure: Lower Third Molar Extraction; Drug: Hyaluronidase
- Placebo (Placebo Comparator): Lower Third Molar Extraction -- Anesthetic: 3.6 mL of the LA 2% HCl mepivacaine with 1:100,000 epinephrine + Placebo (0.9% saline)
  Interventions: Drug: 3.6mL 2% Mepivacaine with 1:100,000 epinephrine; Procedure: Lower Third Molar Extraction; Drug: Placebo

INTERVENTIONS:
Drug: 3.6mL 2% Mepivacaine with 1:100,000 epinephrine — Local anesthetic with vasoconstrictor
  Other Names: Mepivacaine with epinephrine
Procedure: Lower Third Molar Extraction — Lower Third Molar Extraction with LA + hyaluronidase (or placebo)
  Other Names: Molar surgery
Drug: Hyaluronidase — 75RTU Hyaluronidase administration concomitant to the local anesthetic
  Arms: Hyaluronidase
Drug: Placebo — 1mL 0.9% saline administration concomitant to the local anesthetic
  Other Names: Saline; 0.9% NaCl
  Arms: Placebo

SUMMARY:
Among the adjuvants to local anaesthetics (LA), the enzyme hyaluronidase is most often used as a diffuser agent of the LA in ophthalmic anaesthesia. It serves to improve clinical efficacy and prolong anaesthesia as an alternative to long-lasting and potentially more dangerous LA, especially in patients with increased cardiovascular risk. There is scarce clinical data about the safety of the use of hyaluronidase in dental procedures.

This study aimed to compare hemodynamic and electrocardiographic variables during a dental surgical procedure using a local anaesthetic associated with hyaluronidase or placebo in healthy subjects.

DETAILED DESCRIPTION:
This double-blind crossover "split-mouth" trial evaluated the cardiovascular effects induced by 3.6 mL of the LA 2% HCl mepivacaine with 1:100,000 epinephrine, concomitantly with 75 TRU/mL hyaluronidase or placebo in inferior alveolar nerve block, for the performance of bilateral and symmetrical third molar surgery in 20 outpatients. Cardiovascular parameters, including systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate (HR), were monitored using oscillometric and photoplethysmographic methods in 10 clinical stages. Electrocardiographic records (ECG) of 12 leads were obtained in four steps. Hyaluronidase injected concomitantly with LA did not induce changes in SBP, DBP and HR compared to placebo. There were no instances of ST segment depression, ST segment elevation, wide QRS complex extrasystoles, or narrow QRS complex extrasystoles.

To date, few studies in dentistry have investigated the effects of local anaesthetic efficacy in hyaluronidase, and even fewer have studied the relation to systemic effects induced by this interaction.

The use of LA injected concomitantly with 75 TRU/mL of hyaluronidase is safe when using this dose and route of administration.

Clinical Relevance: In dentistry, few studies have investigated the effects of hyaluronidase on local anaesthetic efficacy, and even fewer have examined the possible systemic effects induced by this interaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients should present bilateral lower third molars (teeth 38 and 48) for extraction and identical anatomical arrangement;
* Absence of significant clinical morbidities, ASA I (American Society of Anesthesiologists, 1963);
* Aged over 18 years.

Exclusion Criteria:

* Women during pregnancy or lactation;
* Smokers;
* History of sensitivity to any drug used in the research;
* Presence or history of cancer or an infectious lesion;
* Individuals who used any medication in the last 15 days (except oral contraceptives);
* Presence of abscess or pericoronitis in the region to be operated;
* Patients who required supplemental anaesthesia upon anaesthetic block of the inferior alveolar nerve (post-randomisation exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Arrhythmia | 5min before anaesthesia
  Atrial or ventricular arrhythmias: isolated, paired or clustered extrasystoles, tachycardia, bradycardia and fibrillation.

SECONDARY OUTCOMES:
PR segment | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Duration of the PR segment, in milliseconds.
QRS complex | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Duration of the QRS complex, in milliseconds.
Change from baseline Heart rate | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Change from baseline Heart rate (evaluated period - baseline), in beats per minute. Values will be expressed as the absolute difference and the percentage of change.
Corrected QT | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Duration of the calculated corrected QT segment (QTc) in milliseconds.
Heart rate (absolute values) | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Heart rate, (absolute values) in beats per minute.

OTHER OUTCOMES:
Systolic Pressure (absolute values) | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  Systolic Blood Pressure (absolute values), in mmHg.
Diastolic Pressure (absolute values) | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  Diastolic Blood Pressure, in mmHg.
Mean Blood Pressure (absolute values) | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  Mean Blood Pressure, in mmHg.
Change from baseline Diastolic Pressure | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Change from baseline Diastolic Blood Pressure (evaluated period - baseline), in mmHg. Values will be expressed as the absolute difference and the percentage of change.
Change from baseline Systolic Pressure | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Change from baseline Systolic Blood Pressure (evaluated period - baseline), in mmHg. Values will be expressed as the absolute difference and the percentage of change.
Change from baseline Mean Arterial Blood Pressure | 5min before anaesthesia; During anaesthetic injection; 5min after anaesthesia; Incision; Syndesmotomy; Luxation; Avulsion; Curetage; Suture; 1 hour after the end of surgery (At Patient discharge) and in the 7th postoperative day
  • Change from baseline Mean Arterial Blood Pressure (evaluated period - baseline), in mmHg. Values will be expressed as the absolute difference and the percentage of change.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo F Prado, PhD, Study Chair — FMUSP; Maria A Borsatti, PhD, Study Director — FOUSP; Rodney G Rocha, PhD, Study Director — FOUSP; Helena R Tornelli, MD, S, Study Chair — FOUSP; Renata MS Prado, MS, S, Study Chair — FOUSP
Locations (1):
- Stomatology Department, FOUSP, São Paulo, São Paulo, Brazil